CLINICAL TRIAL: NCT01235221
Title: Open-Label Extension Study to Evaluate the Safety and Tolerability of Oral Fampridine SR in Canadian Subjects With Multiple Sclerosis Who Participated in Acorda Extension Trials
Brief Title: Open Label Extension Study to Evaluate the Safety and Tolerability of Oral Fampridine-Sustained Release (SR) in Canadian Participants With Multiple Sclerosis Who Participated in Acorda Extension Trials.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 218MS301
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — 4-Aminopyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BIIB041 (Fampridine-SR) (Experimental): Participants take 10 mg sustained-release tablets of fampridine twice daily for up to 27 months or until the product is commercially available.
  Interventions: Drug: BIIB041 (Fampridine-SR)

INTERVENTIONS:
Drug: BIIB041 (Fampridine-SR) — 10 mg twice a day (BID) sustained-release (SR) tablets by mouth for up to 27 months (in addition to treatment in previous studies) or until the product is commercially available, whichever comes first. Doses of study treatment must be spaced at least 12 hours apart.
  Other Names: Dalfampridine; Fampridine-ER; Ampyra; Fampyra; Fampridine-PR

SUMMARY:
The primary objective of the study is to evaluate the long-term safety and tolerability of BIIB041 (fampridine-sustained release (SR)) treatment in Canadian participants with multiple sclerosis (MS) who previously participated in the registrational and extension studies conducted by Acorda. Those studies include NCT00654927 (MS-F202EXT), NCT00648908 (MS-F203EXT) and NCT00649792 (MS-F204EXT).

ELIGIBILITY:
Key Inclusion Criteria :

1. Previously enrolled in 1 of the 3 Acorda-sponsored studies (MS-F202EXT, MS-F203EXT, and MS-F204EXT) and continuing to receive fampridine-SR.
2. Willing to comply with the required scheduling and assessments of the protocol.
3. Female subjects of childbearing potential, regardless of sexual activity, must have a negative urine pregnancy test, and must practice effective contraception during the study and be willing and able to continue contraception for 1 month after their last dose of study treatment.

Key Exclusion Criteria:

1. Discontinued prematurely from the preceding study ((MS-F202EXT, MS-F203EXT, or MS-F204EXT).
2. Any prior history of seizure, epilepsy, or other convulsive disorder.
3. Any clinically significant abnormal laboratory values.
4. New history of moderate or severe renal impairment.
5. New history of angina, uncontrolled hypertension, clinically significant cardiac arrhythmias, or any other clinically significant cardiovascular abnormality, as judged by the Investigator.
6. Any significant change in overall health that would preclude subject's participation in the study, in the opinion of the Investigator.
7. Known allergy to pyridine-containing substances or any of the inactive ingredients of the fampridine-SR tablet
8. Received an investigational drug, except fampridine-SR under the preceding study (MS-F202EXT, MS-F203EXT, or MS-F204EXT), within the last 30 days, or the subject is scheduled to enroll in an investigational drug at any time during the study.
9. A history of drug or alcohol abuse within the past year.
10. Treatment with other forms of fampridine or 4-AP (e.g., compounded formulation of 4-AP) or 3,4-diaminopyridine (3,4-DAP).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) and serious adverse events (SAEs) as well as Changes in vital signs and clinical laboratory assessments | From Screening (Day 0) to Termination (Month 27)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (5):
- Canada (5):
  - Foothills Medical Center, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - River Valley Health, Fredericton, New Brunswick
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Ottawa Hospital General Campus, Ottawa, Ontario